CLINICAL TRIAL: NCT05527717
Title: REvaSCUlarization StratEgy of Multivessel Coronary Artery Disease for Patients with Acute Myocardial Infarction Complicated by Cardiogenic SHOCK Undergoing Veno-arterial Extracorporeal Membrane Oxygenator: Randomized-Controlled Trial (RESCUE-SHOCK)
Brief Title: Revascularization Strategy of Multivessel Disease for Patients with Acute Myocardial Infarction Complicated by Cardiogenic Shock Undergoing Veno-arterial Extracorporeal Membrane Oxygenator
Acronym: RESCUE-SHOCK
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeong Hoon Yang, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESCUE-SHOCK
Record Dates: First submitted 2022-08-27; First posted 2022-09-02 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Cardiogenic Shock; Acute Myocardial Infarction; Multi Vessel Coronary Artery Disease; Extracorporeal Membrane Oxygenation
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, two-arm, randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Culprit-lesion only PCI arm (Active Comparator): Patients will receive culprit-lesion only PCI.
  Interventions: Procedure: Culprit lesion only PCI
- Immediate multi-vesesl PCI arm (Experimental): Patients will receive immediate multi-vessel PCI.
  Interventions: Procedure: Immediate multi-vessel PCI

INTERVENTIONS:
Procedure: Culprit lesion only PCI — Randomization will be done after coronary angiography before or during primary PCI for IRA. Patients will be randomized to either immediate multi-vesesl PCI group or culprit-lesion only PCI group with 1:1 ratio.
  This group will be taken culprit-lesion only PCI during primary PCI.
  Arms: Culprit-lesion only PCI arm
Procedure: Immediate multi-vessel PCI — Randomization will be done after coronary angiography before or during primary PCI for IRA. Patients will be randomized to either immediate multi-vesesl PCI group or culprit-lesion only PCI group with 1:1 ratio.
  This group will be taken immediate multi-vesesl PCI during primary PCI.
  Arms: Immediate multi-vesesl PCI arm

SUMMARY:
This study is a prospective, open-label, two-arm, randomized multicenter trial to identify whether immediate multi-vessel PCI would be better in clinical outcomes compared with culprit lesion-only PCI for AMI and multi-vessel disease with an advanced form of CS patients who require veno-arterial extracorporeal membrane oxygenator (VA-ECMO).

DETAILED DESCRIPTION:
Cardiogenic shock (CS) is a fatal complication of acute myocardial infarction (AMI). Until now, in this setting, it has been well-known that early revascularization with percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG) was associated with improved clinical outcomes although the rate of mortality remains still high in the mechanical circulatory support (MCS) era. In real-world practice, since clinically significant non-infarct related artery (non-IRA) stenosis or occlusion in addition to an IRA can be found in 70% to 80% of patients with AMI complicated by CS, the decision of revascularization strategy is a crucial issue to improve clinical outcomes in CS patients with multivessel disease. The 2013 American College of Cardiology (ACC)/American Heart Association (AHA) and the 2017 European Society of Cardiology (ESC) guidelines recommend considering PCI of severe stenosis in non-IRA during a primary procedure to improve overall myocardial perfusion and hemodynamic stability for patients with AMI and CS. However, the CULPRIT-SHOCK trial, which is the largest randomized trial in CS, demonstrated the 30-day risk of a composite of death or severe renal failure leading to renal-replacement therapy was higher in the immediate multi-vessel PCI than in the culprit lesion-only PCI group. In this regard, the recently updated guidelines do not recommend the routine non-IRA revascularization during primary PCI and it should be considered in selected cases in which there is a very severe flow-limiting non-IRA stenosis irrigating a large myocardial area. Nevertheless, there is still some unsolved issue regarding the role of non-IRA revascularization in AMI patients with CS. Majority of enrolled patients in the CULPRIT-SHOCK trial might have a mild form of CS (median systolic blood pressure of 100) and few patients received MCS devices (28.3% of study population). Furthermore, the mortality benefits of culprit-only PCI were attenuated at 1-year follow-up with an increased risk of repeat revascularization and hospitalization for heart failure. In contrast to the CULPRIT-SHOCK trial, the recent large United State registry from National Cardiovascular Data Registry demonstrated that the benefits of multi-vessel PCI in patients with non-ST-segment elevation MI and CS was more pronounced in those requiring MCS. In addition, recent data from the Korea Acute Myocardial Infarction National Health Registry showed that multivessel PCI was associated with a lower risk of all-cause death than culprit-only PCI, suggesting possible benefit of nonculprit lesion revascularization during the index hospitalization on long-term clinical outcomes.

Therefore, the current randomized trial sought to identify whether immediate multi-vessel PCI would be better in clinical outcomes compared with culprit lesion-only PCI for AMI and multi-vessel disease with advanced form of CS patients who requiring veno-arterial extracorporeal membrane oxygenator (VA-ECMO).

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 19 years of age
* Patients presented with AMI (ST-segment elevation MI [STEMI] or non-ST-segment elevation MI [NSTEMI]) complicated by CS (SCAI Shock classification C, D or E) who requiring VA-ECMO.
* Target lesions amenable for planned primary PCI by operators' decision
* Patients with multi-vessel disease

Exclusion Criteria:

* Other causes of shock (hypovolemia, sepsis, obstructive shock).
* Shock due to mechanical complication to MI (rupture of papillary muscle, the ventricular septum, or free wall).
* Unwitnessed out of hospital cardiac arrest with persistent Glasgow coma scale <8 after the return of spontaneous circulation.
* Patients with single-vessel disease (Patients with single-vessel disease will be enrolled in the RESCUE-SHOCK registry)
* Onset of shock >24 hours.
* Known heparin intolerance.
* Other severe concomitant disease with limited life expectancy < 6 months
* Pregnancy or breast feeding
* Do not resuscitate wish

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2022-11-16 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Rates of all-cause mortality or advanced heart failure requiring cardiac replacement therapy | 90 days after primary PCI
  all-cause mortality or requiring left ventricular assisted device (LVAD) insertion or heart transplantation)

SECONDARY OUTCOMES:
Rates of In-hospital mortality | Up to 30 days
  Death by any cause in hospital
Rates of In-hospital cardiac mortality | Up to 30 days
  Death by cardiac cause in hospital
Rates of VA-ECMO weaning success | Up to 30 days
  Successful weaning of VA-ECMO was defined as successful removal of VA-ECMO and not requiring further mechanical support because of recurring cardiogenic shock over the following 48 hours.
Time to VA-ECMO weaning | Up to 30 days
  Time from VA-ECMO insertion to VA-ECMO weaning
Rates of critical limb ischemia after successful VA-ECMO weaning | Up to 30 days
  Critical limb ischemia is defined as limb pain that occurs at rest, or impending limb loss that is caused by severe compromise of blood flow to the affected extremity. (Rutherford classification 4, 5, or 6)
Cerebral Performance Category (CPC) 3-5 at discharge | Up to 30 days
  Neurologic performance scale at discharge
Length of intensive-care unit (ICU) stay | Up to 30 days
  ICU stay day
Total procedural time | Immediate after the index procedure
  Procedural time (minutes)
Total amount of contrast use | Immediate after the index procedure
  Contrast use (cc)
Rates of all-cause mortality | 90 Days and 12 months after primary PCI
  Death by any cause
Rates of cardiac mortality | 90 Days and 12 months after primary PCI
  Death by cardiac cause
Requirement of cardiac replacement therapy | 90 Days and 12 months after primary PCI
  LVAD insertion or heart transplantation
Requirement of renal replacement therapy | 90 Days and 12 months after primary PCI
  Continuous renal replacement therapy, hemodialysis, or peritoneal dialysis
Rates of myocardial infarction (MI) | 90 Days and 12 months after primary PCI
  spontaneous MI during follow-up
Rates of MI related to culprit vessel | 90 Days and 12 months after primary PCI
  MI related to culprit vessel during follow-up
Rates of MI related to non-culprit vessel | 90 Days and 12 months after primary PCI
  MI related to non-culprit vessel during follow-up
Rates of stent thrombosis | 90 Days and 12 months after primary PCI
  Academic Research Consortium (ARC)-defined definite or probable stent thrombosis
Rates of Re-hospitalization due to heart failure | 90 Days and 12 months after primary PCI
  Re-hospitalization due to heart failure during follow-up
Rates of Re-hospitalization due to any cause | 90 Days and 12 months after primary PCI
  Re-hospitalization due to any cause during follow-up
Rates of target-lesion revascularization (TLR) | 90 Days and 12 months after primary PCI
  TLR during follow-up
Rates of target-vessel revascularization (TVR) | 90 Days and 12 months after primary PCI
  TVR during follow-up
Rates of repeat revascularization | 90 Days and 12 months after primary PCI
  Repeat revascularization during follow-up
Rates of cerebrovascular accident | 90 Days and 12 months after primary PCI
  Cerebrovascular accident during follow-up
Rates of bleeding | 90 Days and 12 months after primary PCI
  Bleeding ARC [BARC] type 2, 3, or 5
Rates of major bleeding | 90 Days and 12 months after primary PCI
  (BARC type 3 or 5

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Hoon Yang, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No